CLINICAL TRIAL: NCT05307900
Title: Ultrasonography Confirmation of Feeding Tube Placement in Critically Ill Patients
Brief Title: Ultrasonography Confirmation of Feeding Tube Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Rufinah Teo, Lecturer and Consultant Anesthesiologist , Department of Anesthesia and Intensive Care, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FF-2020-505
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Feeding Tube
Keywords: ultrasonography; ryle's tube

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients requiring intubations (Experimental): All intubated patients with feeding tube
  Interventions: Other: Confirmation of feeding tube placement in critically ill patients

INTERVENTIONS:
Other: Confirmation of feeding tube placement in critically ill patients — Confirmation of feeding tube placement using ultrasonography

SUMMARY:
To compare the correct placement of feeding tube in critically ill patients in ICU using ultrasonography versus chest radiography

DETAILED DESCRIPTION:
Patients who are indicated for feeding tube (FT) placement in ICU will be recruited in this study. Written informed consent will be obtained from next of kin.

Feeding tubes will be inserted by ICU oncall anaesthesiologist as per protocol. The FTof polyvinyl chloride with calibre of 12-16 French will be used. The Nose-Ear-Xiphoid method will be used to measure the tube insertion distance, adding the distance from tip of the patient's nose to the earlobe and from the earlobe to the xiphoid. The tip of tube lubricated prior to insertion in all cases. Orogastric tube placement will be done if nasal route placement is unsuccessful or contraindicated.

Once the correct placement is confirmed by auscultation and aspirate method, the tube will be secured to patient's nose with adhesive tape. For the purpose of this study, verification of tube placement will be done with bedside ultrasound prior to X-ray.

Ultrasound verification of tube placement will be done by a single investigator who received training on oesophageal and gastric ultrasound from radiologist. 'Sonosite SII' (by Fujifilm Sonosite, Inc) ultrasound machine will be used to conduct this study. A linear probe (L38xi, 10-5MHz) will be placed transversely at the anterior neck and focused on visible part of oesophagus which will be just below the left thyroid lobe. A curved probe (C35x, 8-3MHz) will be placed at subxiphoid area orientated towards left upper abdominal quadrant to visualize the stomach and by angulating the probe towards the left subcostal area, the gastric body can be identified in transversal plane just beside the left lobe of liver as internal landmark.

The ultrasound examination will be considered positive if the FT visualized as a hyperechogenic circle posterior to left thyroid lobe adjacent to trachea, and as a hyperechogenic point in the stomach. If the FT seen in the oesophagus and not in stomach, a 20mls of air will be injected through the FT using pine tip syringe while observing dynamic fogging in the stomach. FT is considered in the gastric body in the presence of fogging. Total duration of ultrasound confirmation of FT will be recorded. Following completion of ultrasound confirmation of FT, a chest x-ray will be done for all the patients as per usual. The chest x-ray will be reviewed by ICU team who are blinded from this study.

Dichotomous results either positive or negative of ultrasound examination and x-ray evaluation will be obtained. The criteria for confirmation of FT via ultrasonography will be the positive neck scan and either positive subxiphoid scan or positive fogging test. The ICU oncall anaesthesiologist will be informed immediately in the event of suspected FD misplacement (negative neck scan, negative subxiphoid scan and negative fogging) and an urgent chest x-ray will be requested. Additional data such as duration of ultrasound examination (procedure time) will be included in this study.

ELIGIBILITY:
Inclusion Criteria:

All the patients, aged > 18 years old that admitting to ICU who require feeding tube insertion

Exclusion Criteria:

1. Any contraindications for FT insertion. e.g. coagulopathy, oesophageal varices
2. History or post gastric by-pass surgeries
3. Known history of nasopharyngeal, oesophagus or stomach carcinoma
4. Neck trauma/swelling including goitre
5. Open wounds at neck or epigastric regions
6. Pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
To compare the correct placement of feeding tube in critically ill patients in ICU using ultrasonography versus chest radiography | 1 year
  Numbers of positive ultrasound verifications of correct placement of feeding tube

SECONDARY OUTCOMES:
To study time taken to perform USG examination to confirm feeding tube placement in critically ill patients | 1 year
  Total duration of ultrasound examination to verify correct placement of feeding tube

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz,, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gok F, Kilicaslan A, Yosunkaya A. Ultrasound-guided nasogastric feeding tube placement in critical care patients. Nutr Clin Pract. 2015 Apr;30(2):257-60. doi: 10.1177/0884533614567714. Epub 2015 Jan 23. PMID 25616518
- [Result] Kim HM, So BH, Jeong WJ, Choi SM, Park KN. The effectiveness of ultrasonography in verifying the placement of a nasogastric tube in patients with low consciousness at an emergency center. Scand J Trauma Resusc Emerg Med. 2012 Jun 12;20:38. doi: 10.1186/1757-7241-20-38. PMID 22691418
- [Result] Yildirim C, Coskun S, Gokhan S, Pamukcu Gunaydin G, Ozhasenekler A, Ozkula U. Verifying the Placement of Nasogastric Tubes at an Emergency Center: Comparison of Ultrasound with Chest Radiograph. Emerg Med Int. 2018 Dec 18;2018:2370426. doi: 10.1155/2018/2370426. eCollection 2018. PMID 30662772
- [Result] Vigneau C, Baudel JL, Guidet B, Offenstadt G, Maury E. Sonography as an alternative to radiography for nasogastric feeding tube location. Intensive Care Med. 2005 Nov;31(11):1570-2. doi: 10.1007/s00134-005-2791-1. Epub 2005 Sep 20. PMID 16172849
- [Result] Chenaitia H, Brun PM, Querellou E, Leyral J, Bessereau J, Aime C, Bouaziz R, Georges A, Louis F; WINFOCUS (World Interactive Network Focused On Critical Ultrasound) Group France. Ultrasound to confirm gastric tube placement in prehospital management. Resuscitation. 2012 Apr;83(4):447-51. doi: 10.1016/j.resuscitation.2011.11.035. Epub 2011 Dec 29. PMID 22209831